CLINICAL TRIAL: NCT02749773
Title: Is There a Difference in Oocyte Quality? A Comparison of Two Aspiration Needle Gauges
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HYMC-0026-16
Record Dates: First submitted 2016-04-06; First posted 2016-04-25 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oocyte aspiration with 17G needle (Active Comparator): Oocyte Aspiration with 17G needle.
  Interventions: Device: Oocyte Aspiration needle
- Oocyte aspiration with (20-17G) needle (Active Comparator): Oocyte Aspiration (20-17G) needle.
  Interventions: Device: Oocyte Aspiration needle

INTERVENTIONS:
Device: Oocyte Aspiration needle — Oocyte aspiration in women go through an IVF procedure,.

SUMMARY:
The aim of this study is to determine whether different needle gauges influences the quality of the aspirated oocytes during in-vivo fertilization (IVF).

ELIGIBILITY:
Inclusion Criteria:

* Fertility treatment
* Antral follicle count

Exclusion Criteria:

* Women who refuse to participate

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Oocyte Quality microscopic description. | One year
  Aspirated oocytes from both needle gauges will be compared for quality according to 5 parameters: Polar body, Zona pellucida, Dark cytoplasm, Perivitelline space and Vacuoles.

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Atzmon, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atzmon Y, Michaeli M, Aslih N, Ruzov O, Rotfarb N, Shoshan-Karchovsky E, Shalom-Paz E. Degenerative Oocytes in the Aspirated Cohort Are Not Due to the Aspirating Needle: a Prospective Randomized Pilot Study with Sibling Oocytes. Reprod Sci. 2021 Jul;28(7):1882-1889. doi: 10.1007/s43032-020-00384-3. Epub 2020 Nov 10. PMID 33171516